CLINICAL TRIAL: NCT00867880
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Dose, Crossover Study of the Pharmacokinetics, Safety and Tolerability of Ibuprofen Inejction (IVIb) In Healthy Adult Volunteers
Brief Title: Pharmacokinetic Study Of Ibuprofen Injection (IVIb) In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CPI-CL-011
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: To evaluate the Pharmacokinetic Profile of IVIb

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: IVIb
- 2 (Active Comparator)
  Interventions: Drug: IVIb

INTERVENTIONS:
Drug: IVIb — 800mg IVIb diluted in 200mL NS will be given IV (in the vein) concurrently with an oral placebo on Day 1 and 200ml Normal Saline will be given IV (in the vein)concurrently with 800mg oral ibuprofen on Day 8

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetic profile of a single dose of IVIb administered over 5-7 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 18 and 65 years (at the time of consent).

Exclusion Criteria:

* Participants lacking good venous access in both arms.
* History of allergy or hypersensitivity to NSAIDs or any component of intravenous ibuprofen.
* Have never taken aspirin or ibuprofen
* History of abuse of alcohol or other drugs in the 2 months before CTM administration.
* Have used prescription drugs (not including oral contraceptives) within 14 days before CTM administration or have used aspirin within one week before CTM administration or over-the-counter pain relievers (NSAIDs or acetaminophen) within 3 days before CTM administration.
* Have taken investigational drugs within 30 days before CTM administration.
* Have donated blood or blood products within 30 days before CTM administration.
* Be pregnant or nursing.
* Have had breast cancer.
* Have a clinically significant laboratory test
* Presence or history of the following conditions: asthma, bleeding tendency, hypertension, heart failure, peptic ulcer disease, inflammatory bowel disease, or any other gastrointestinal disorder, renal or hepatic disease..
* Have a calculated creatinine clearance (estimated by means of the Cockcroft-Gault equation) of < 75mL/min
* Inability to understand the requirements of the study. Participants must be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions.
* Refusal to provide written authorization for use and disclosure of protected health information
* Be otherwise unsuitable for the study, in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic profile of a single dose of IVIb administered over 5-7 minutes. | 12 hours

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of a single dose of IVIb in healthy adult participants. | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert Milne, Associate Professor, Principal Investigator — Centre for Pharmaceutical Research
Locations (1):
- Centre for Pharmaceutical Research, Underdale, South Australia, Australia